CLINICAL TRIAL: NCT04799691
Title: Comparison of 2 Ventilatory Support Strategies in Patients With Covid-19 Pneumonia Admitted in ICU : Retrospective Monocentric Study
Brief Title: Comparison of 2 Ventilatory Support Strategies During Coronavirus Disease 2019 (Covid-19) Pneumonia
Acronym: STRATIC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-CHITS-004
Record Dates: First submitted 2021-03-15; First posted 2021-03-16 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
Keywords: Invasive strategy; Non-invasive strategy; Continuous Positive Airway Pressure; High Flow Nasal Canula; Prone position
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Invasive strategy group: Patients admitted in ICU with Covid-19 related pneumonia during COVID19 first period.
  Interventions: Procedure: Invasive ventilation strategy
- Non-invasive strategy group: Patients admitted in ICU with Covid-19 related pneumonia during COVID19 second period.
  Interventions: Procedure: Non-invasive ventilation strategies

INTERVENTIONS:
Procedure: Invasive ventilation strategy — Use of an invasive ventilatory support strategy
  Groups: Invasive strategy group
Procedure: Non-invasive ventilation strategies — Use of non-invasive ventilatory support strategies
  Groups: Non-invasive strategy group

SUMMARY:
This retrospective monocentric study compares 2 ventilatory support strategies on outcomes (length of stay, intubation, mortality) in patients admitted in Intensive Care Unit with Covid-19 related pneumonia : invasive strategy used during the first period and non-invasive strategies (Continuous Positive Airway Pressure, High Flow Nasal Canula, Prone Position) used during the second period.

ELIGIBILITY:
Inclusion Criteria:

* Patient with confirmed SARS COV2 infection
* Acute Respiratory Distress Syndrome
* Patient more than 18 year old

Exclusion Criteria:

* Intensive Care Unit admission for extra pulmonary failure
* "Do Not Reanimated" order
* Patient from another Intensive Care Unit
* Patient objection
* Judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COVID 19 acute hypoxemic respiratory failure admitted in Hospital Sainte Musse ICU in 2020
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Length of stay in ICU | At the moment of ICU discharge or death, up to 3 month
  Number of days spent in ICU

SECONDARY OUTCOMES:
Mortality | At the moment of ICU discharge or death, up to 3 month
  Rate of patients alive at the moment of intensive care unit discharge
Complications | At the moment of ICU discharge or death, up to 3 month
  Number of complications during intensive care unit stay

CONTACTS AND LOCATIONS:
Overall Officials: Aude Garnero, MD, Study Director — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer
Locations (1):
- Hôpital Sainte Musse, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No